CLINICAL TRIAL: NCT05901688
Title: Umbilical Cord Abnormalities in the Prediction of Adverse Pregnancy Outcomes
Acronym: ULOOP
Status: Recruiting | Type: Observational
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Ranjit Akolekar, Consultant in Fetal Medicine & Obstetrics, Medway NHS Foundation Trust
Other Study IDs: 001
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Small for Gestational Age at Delivery; Hypoxic-Ischemic Encephalopathy; Stillbirth; Admission to Neonatal Unit
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Stillbirth | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unselected population: Routine unselected populations at 20-22 weeks and 35-37 weeks
  Interventions: Other: Umbilical cord measurements & observations
- High risk population: High-risk pregnancies attending the placental disorders clinic which have been deemed to be at risk of having adverse pregnancy outcomes.
  Interventions: Other: Umbilical cord measurements & observations

INTERVENTIONS:
Other: Umbilical cord measurements & observations — In the screening study of an unselected population at 20-22 weeks' and 35-37 weeks' gestation, women are offered an ultrasound scan as part of standard care and will be invited to take part in the study which will involve taking the following additional ultrasound measurements:
  1. Umbilical cord coiling index (UCI)
  2. Transverse diameter of umbilical cord (UC)
  3. Transverse diameter of umbilical vein (UV) and artery (UA)
  4. Umbilical vein (UV) Doppler flow characteristics
  5. Presence of nuchal cord

SUMMARY:
The objective of our study is to investigate the association of umbilical cord abnormalities with adverse pregnancy outcomes. The umbilical cord parameters that will be investigated as part of this study include the umbilical cord coiling index (UCI), umbilical cord (UC) diameter, umbilical vein (UV) diameter, UV flow velocity and the presence of nuchal cord. The UCI, UC, UV diameter & flow and presence of nuchal cord will be measured in routine unselected populations at 20-22 weeks and 35-37 weeks gestation during the study period. We will also measure the UC and UV diameter in a nested population of high-risk pregnancies attending our placental disorders clinic which have been deemed to be at risk of having adverse pregnancy outcomes.

Primary objective:

To investigate if prenatal assessment of UCI, UC, UV diameter & flow and presence of nuchal cord measured routinely in unselected screened populations at 20-22 weeks and 35-37 weeks' can provide an independent prediction of pregnancies that develop adverse pregnancy outcomes.

Secondary objectives:

To assess the correlation of UC and UV diameter measured by ultrasound scan and fetal magnetic resonance imaging in prediction of pregnancy outcome. To examine the association of these umbilical cord measurements and observations in a nested cohort of pregnancies in the high-risk placental disorders clinic.

DETAILED DESCRIPTION:
The umbilical diameter is less than 2 cm, grows to a length of 50-60 cm by 28 weeks gestation and contains around 40 helical turns, which are twisted to the left rather than right because of the arrangement of helical muscle fibers in the vessels of the umbilical cord. These twists in the umbilical cord add to the strength of the cord by providing protection and resistance against compression of umbilical vessels. The overall final length of the UC and the number of coils is thought to be determined by the tensile forces due to fetal movements, rate of growth of UA and UV, fetal hemodynamics, distribution of the muscle fibers in the UA and amniotic fluid volume.

One of the common causes of fetal and neonatal adverse outcomes such as stillbirths or hypoxic ischaemic encephalopathy (HIE) is fetal hypoxia. The optimally oxygenated blood is transferred from the maternal blood to the fetus, crossing the placenta and the UC to reach fetal circulation. There are several studies which demonstrate that fetal hypoxia due to placental causes, whether chronic or acute, can lead to reduced transfer of oxygen and nutrition to the fetus. There is evidence from clinical and histological studies that impaired trophoblastic proliferation causes impaired placentation and leads to reduced oxygen transfer to the fetus resulting in preeclampsia (PE), fetal growth restriction (FGR) or stillbirth. However, there is limited and uncertain evidence regarding the contribution of UC abnormalities in the prediction of pregnancies with fetal hypoxia that result in hypoxic adverse outcomes such as HIE and stillbirth. There is need for further research to investigate the causes related to UC as not all hypoxic adverse outcomes have a placental etiology and a significant proportion of pregnancies with FGR, stillbirth and HIE have no ultrasound or histological evidence of impaired placentation, suggesting that there may be other factors in addition to the placenta that lead to such hypoxic morbidity.

There are studies published in literature demonstrating an association between UC abnormalities and adverse pregnancy outcomes such as FGR, PE, stillbirth or adverse outcomes such as caesarean section (CS) for fetal distress; but many of these are postnatal studies based on morphological and histological examination rather than prospective cohort studies carried out in the antenatal period. The few studies that investigate UC abnormalities in prenatal period are retrospective case-control studies with a relatively small sample size. This makes the findings less generalizable and overall difficult to effectively assess the precise contribution of UC abnormalities detected on ultrasound in the prenatal period that can potentially improve management and prevent such adverse outcomes.

This is a prospective observational cohort study carried out at a single center. This study will be conducted in compliance with the study protocol, the Declaration of Helsinki (1996), the principles of Good Clinical Practice (GCP) and applicable regulatory requirements. The study will be reviewed and approved by the Research Ethics Committees (REC) and competent authorities.

At our centre, all women booked for their maternity care are offered 3 routine ultrasound scans in their pregnancy: 11-13 weeks', 20-22 weeks' and at 35-37 weeks' gestation. Pregnancies that are deemed to be at high risk for delivery of a small for gestational age neonate are referred to a specialist placental disorders clinic for closer antenatal monitoring and fetal surveillance. At these visits, we ensure that there is a complete record of their personal, medical and obstetric history and perform an ultrasound scan to assess fetal growth, amniotic fluid and Doppler studies. This prospective study has two parts: first, a prospective observational cohort study in an unselected population and a nested cohort study in a high-risk population. Those agreeing to take part will be offered a patient information sheet and requested to sign a consent form, confirming their willingness to participate.

Prospective cohort study: In the screening study of an unselected population at 20-22 weeks' and 35-37 weeks' gestation, women are offered an ultrasound scan as part of standard care and will be invited to take part in the study which will involve taking the following additional ultrasound measurements:

1. Umbilical cord coiling index (UCI)
2. Transverse diameter of umbilical cord (UC)
3. Transverse diameter of umbilical vein (UV) and artery (UA)
4. Umbilical vein (UV) Doppler flow characteristics
5. Presence of nuchal cord

Nested cohort study: In the nested cohort study of the high-risk pregnancies, women are offered measurement of fetal biometry and Doppler assessments including UA Doppler as part of the standard care. Women will be invited to take part in the study which will involve taking the following additional ultrasound measurements:

1. Umbilical cord coiling index (UCI)
2. Transverse diameter of umbilical cord (UC)
3. Transverse diameter of umbilical vein (UV) and artery (UA)
4. Umbilical vein (UV) Doppler flow characteristics

The additional measurements of UC, UV and nuchal cord will only add 2-3 minutes of examination time and will not affect the care of women attending for their routine assessments as well as in the high-risk placental disorders clinic. These measurements taken as part of the study will not be available for clinical management and will be analysed after the completion of the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancies.
2. Women booked at our unit prior to 20 weeks' gestation.

Exclusion Criteria:

1. Multiple pregnancies.
2. Age < 16 years.
3. Those unable to provide consent.
4. Pregnancies with fetal abnormalities.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Gender eligibility based on biological gender
Study Population: The study will be carried out in two cohorts: the first is the cohort of unselected population of pregnancies attending for their routine pregnancy care and ultrasound appointments at 20-22 weeks and 35-37 weeks. A nested cohort study will also be carried out in a high-risk cohort of pregnancies referred to the placental disorders clinic for women who have risk factors for delivering a small for gestational age baby or those at risk of developing preeclampsia.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Delivery of small for gestational age (SGA) neonate | 2 years
  Birth weight below the 5th and 10th percentile
Emergency CS for fetal distress | 2 years
  Caesarean section carried out for fetal heart rate abnormalities in labour
Hypoxic ischaemic encephalopathy | 2 years
  Brain damage in neonates causes due to lack of oxygen and confirmed on ultrasound scan
Stillbirth | 2 years
  Death of a fetuses between 24 weeks and before the birth of the baby
Composite hypoxic morbidity | 2 years
  A composite outcome measures of any of the above outcome measures

SECONDARY OUTCOMES:
Preterm delivery < 37 weeks | 2 years
  Spontaneous and iatrogenic preterm delivery
Development of preeclampsia | 2 years
  High blood pressure developing in pregnancy based on ISSHP criteria
Admission to neonatal intensive care unit | 2 years
  Admission to intensive or high-dependency care

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit Akolekar, MD MRCOG PhD, Principal Investigator — Medway NHS Foundation Trust
Locations (1):
- Medway NHS Foundation Trust, Gillingham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hegazy AA. Anatomy and embryology of umbilicus in newborns: a review and clinical correlations. Front Med. 2016 Sep;10(3):271-7. doi: 10.1007/s11684-016-0457-8. Epub 2016 Sep 7. PMID 27473223
- [Background] Moshiri M, Zaidi SF, Robinson TJ, Bhargava P, Siebert JR, Dubinsky TJ, Katz DS. Comprehensive imaging review of abnormalities of the umbilical cord. Radiographics. 2014 Jan-Feb;34(1):179-96. doi: 10.1148/rg.341125127. PMID 24428290
- [Background] Mitchell KE, Weiss ML, Mitchell BM, Martin P, Davis D, Morales L, Helwig B, Beerenstrauch M, Abou-Easa K, Hildreth T, Troyer D, Medicetty S. Matrix cells from Wharton's jelly form neurons and glia. Stem Cells. 2003;21(1):50-60. doi: 10.1634/stemcells.21-1-50. PMID 12529551
- [Background] Pacora P, Romero R, Jaiman S, Erez O, Bhatti G, Panaitescu B, Benshalom-Tirosh N, Jung EJ, Hsu CD, Hassan SS, Yeo L, Kadar N. Mechanisms of death in structurally normal stillbirths. J Perinat Med. 2019 Feb 25;47(2):222-240. doi: 10.1515/jpm-2018-0216. PMID 30231013
- [Background] Man J, Hutchinson JC, Heazell AE, Ashworth M, Jeffrey I, Sebire NJ. Stillbirth and intrauterine fetal death: role of routine histopathological placental findings to determine cause of death. Ultrasound Obstet Gynecol. 2016 Nov;48(5):579-584. doi: 10.1002/uog.16019. Epub 2016 Oct 25. PMID 27781319
- [Background] Ashoor G, Syngelaki A, Papastefanou I, Nicolaides KH, Akolekar R. Development and validation of model for prediction of placental dysfunction-related stillbirth from maternal factors, fetal weight and uterine artery Doppler at mid-gestation. Ultrasound Obstet Gynecol. 2022 Jan;59(1):61-68. doi: 10.1002/uog.24795. PMID 34643306
- [Background] Hammad IA, Blue NR, Allshouse AA, Silver RM, Gibbins KJ, Page JM, Goldenberg RL, Reddy UM, Saade GR, Dudley DJ, Thorsten VR, Conway DL, Pinar H, Pysher TJ; NICHD Stillbirth Collaborative Research Network Group. Umbilical Cord Abnormalities and Stillbirth. Obstet Gynecol. 2020 Mar;135(3):644-652. doi: 10.1097/AOG.0000000000003676. PMID 32028503
- [Background] Akolekar R, Tokunaka M, Ortega N, Syngelaki A, Nicolaides KH. Prediction of stillbirth from maternal factors, fetal biometry and uterine artery Doppler at 19-24 weeks. Ultrasound Obstet Gynecol. 2016 Nov;48(5):624-630. doi: 10.1002/uog.17295. PMID 27854387
- [Background] Tantbirojn P, Saleemuddin A, Sirois K, Crum CP, Boyd TK, Tworoger S, Parast MM. Gross abnormalities of the umbilical cord: related placental histology and clinical significance. Placenta. 2009 Dec;30(12):1083-8. doi: 10.1016/j.placenta.2009.09.005. Epub 2009 Oct 22. PMID 19853300
- [Background] Jessop FA, Lees CC, Pathak S, Hook CE, Sebire NJ. Umbilical cord coiling: clinical outcomes in an unselected population and systematic review. Virchows Arch. 2014 Jan;464(1):105-12. doi: 10.1007/s00428-013-1513-2. Epub 2013 Nov 21. PMID 24259031
- [Background] Damasceno EB, de Lima PP. Wharton's jelly absence: a possible cause of stillbirth. Autops Case Rep. 2013 Dec 31;3(4):43-47. doi: 10.4322/acr.2013.038. eCollection 2013 Oct-Dec. PMID 28584806
- [Background] de Laat MW, Franx A, van Alderen ED, Nikkels PG, Visser GH. The umbilical coiling index, a review of the literature. J Matern Fetal Neonatal Med. 2005 Feb;17(2):93-100. doi: 10.1080/14767050400028899. PMID 16076615
- [Background] de Laat MW, van Alderen ED, Franx A, Visser GH, Bots ML, Nikkels PG. The umbilical coiling index in complicated pregnancy. Eur J Obstet Gynecol Reprod Biol. 2007 Jan;130(1):66-72. doi: 10.1016/j.ejogrb.2006.01.018. Epub 2006 Mar 2. PMID 16513244
- [Background] Strong TH Jr, Jarles DL, Vega JS, Feldman DB. The umbilical coiling index. Am J Obstet Gynecol. 1994 Jan;170(1 Pt 1):29-32. PMID 8296839
- [Background] De Laat MW, Franx A, Nikkels PG, Visser GH. Prenatal ultrasonographic prediction of the umbilical coiling index at birth and adverse pregnancy outcome. Ultrasound Obstet Gynecol. 2006 Oct;28(5):704-9. doi: 10.1002/uog.2786. PMID 16952204
- [Background] El Behery MM, Nouh AA, Alanwar AM, Diab AE. Effect of umbilical vein blood flow on perinatal outcome of fetuses with lean and/or hypo-coiled umbilical cord. Arch Gynecol Obstet. 2011 Jan;283(1):53-8. doi: 10.1007/s00404-009-1272-0. Epub 2009 Nov 7. PMID 19898858
- [Background] Degani S, Leibovich Z, Shapiro I, Gonen R, Ohel G. Early second-trimester low umbilical coiling index predicts small-for-gestational-age fetuses. J Ultrasound Med. 2001 Nov;20(11):1183-8. doi: 10.7863/jum.2001.20.11.1183. PMID 11758023
- [Background] Jo YS, Jang DK, Lee G. The sonographic umbilical cord coiling in late second trimester of gestation and perinatal outcomes. Int J Med Sci. 2011;8(7):594-8. doi: 10.7150/ijms.8.594. Epub 2011 Oct 7. PMID 22022212
- [Background] Sharma B, Bhardwaj N, Gupta S, Gupta PK, Verma A, Malviya K. Association of umbilical coiling index by colour Doppler ultrasonography at 18-22 weeks of gestation and perinatal outcome. J Obstet Gynaecol India. 2012 Dec;62(6):650-4. doi: 10.1007/s13224-012-0230-0. Epub 2012 Aug 17. PMID 24293842
- [Background] Mittal A, Nanda S, Sen J. Antenatal umbilical coiling index as a predictor of perinatal outcome. Arch Gynecol Obstet. 2015 Apr;291(4):763-8. doi: 10.1007/s00404-014-3456-5. Epub 2014 Sep 11. PMID 25209352
- [Background] Kosus A, Kosus N, Turhan NO. Is there any relation between umbilical artery and vein diameter and estimated fetal weight in healthy pregnant women? J Med Ultrason (2001). 2012 Oct;39(4):227-34. doi: 10.1007/s10396-012-0360-0. Epub 2012 May 9. PMID 27279109
- [Background] Tutus S, Asal N, Uysal G, Sahin H. Is there a relationship between high birth weight and umbilical vein diameter? J Matern Fetal Neonatal Med. 2021 Nov;34(21):3609-3613. doi: 10.1080/14767058.2020.1814247. Epub 2020 Oct 20. PMID 33081536
- [Background] Di Naro E, Raio L, Ghezzi F, Franchi M, Romano F, Addario VD. Longitudinal umbilical vein blood flow changes in normal and growth-retarded fetuses. Acta Obstet Gynecol Scand. 2002 Jun;81(6):527-33. PMID 12047306
- [Background] Clapp JF 3rd, Stepanchak W, Hashimoto K, Ehrenberg H, Lopez B. The natural history of antenatal nuchal cords. Am J Obstet Gynecol. 2003 Aug;189(2):488-93. doi: 10.1067/s0002-9378(03)00371-5. PMID 14520223
- [Background] Hayes DJL, Warland J, Parast MM, Bendon RW, Hasegawa J, Banks J, Clapham L, Heazell AEP. Umbilical cord characteristics and their association with adverse pregnancy outcomes: A systematic review and meta-analysis. PLoS One. 2020 Sep 24;15(9):e0239630. doi: 10.1371/journal.pone.0239630. eCollection 2020. PMID 32970750